CLINICAL TRIAL: NCT00733655
Title: Histological Samples From Patients With Hereditary Haemorrhagic Telangiectasia
Brief Title: Study of Histological Samples From Patients With Hereditary Haemorrhagic Telangiectasia
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: IC/CLS5
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Histological samples

SUMMARY:
In this study the investigators will obtain histological samples from people with hereditary haemorrhagic telangiectasia (HHT, also known as Osler-Weber-Rendu Syndrome).

DETAILED DESCRIPTION:
HHT is an inherited condition that leads to the development of dilated and fragile blood vessels. We propose to obtain small skin samples from patients with HHT in order to analyze the samples using histological methods, and study the properties of vascular endothelial cells derived from patients. We hypothesize that these cells will show differences when compared to normal endothelial cells, which may be confirmed in single time point analyses in histological samples. We anticipate that that these findings may help to explain aspects of the HHT disease phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Hereditary Haemorrhagic Telangiectasia

Exclusion Criteria:

* Unable to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hereditary hemorrhagic telangiectasia (HHT)
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2008-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire L Shovlin, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Hammersmith Campus, London, United Kingdom

REFERENCES:
- [Result] Shovlin CL, Gilson C, Busbridge M, Patel D, Shi C, Dina R, Abdulla FN, Awan I. Can Iron Treatments Aggravate Epistaxis in Some Patients With Hereditary Hemorrhagic Telangiectasia? Laryngoscope. 2016 Nov;126(11):2468-2474. doi: 10.1002/lary.25959. Epub 2016 Apr 23. PMID 27107394